CLINICAL TRIAL: NCT06271018
Title: Prospective, Observational Study Assessing Safety and Efficacy of Biosimilar of Tocilizumab in Giant Cell Arteritis (GCA) With Active Aortitis
Brief Title: TocILizumab in aorTitis in GCA (TILT)
Acronym: TILT
Status: Recruiting | Type: Observational
Sponsor: Groupe français d'étude des Maladies Inflammatoires de loeil (Other)
Responsible Party: Sponsor
Other Study IDs: GMIO-2024-0001
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Aortitis; Giant Cell Arteritis (GCA)
Keywords: Giant Cell Arteritis (GCA); Aortitis; Tocilizumab
MeSH Terms: conditions — Aortitis; Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aortitis in GCA: Adult patients with active aortitis associated with GCA, requiring treatment with Tocilizumab biosimilar used within the scope of its market authorization (standard of care)

SUMMARY:
This is a french multicenter observational study assessing safety and efficacy of biosimilar of Tocilizumab in Giant Cell Arteritis (GCA) with active aortitis, including 14 reference centers from the Groupe d'Etude Français des vascularites des gros vaisseaux (GEFA).

Giant Cell Arteritis (GCA), formerly known as temporal arteritis, is the most common form of systemic vasculitis in patients aged ≥ 50 years. GCA is defined by granulomatous arteritis that affects large#sized and medium#sized blood vessels with a predisposition to affect the cranial arteries. Aortitis accounted for more than 50% of GCA patients with the new imaging techniques. Aortitis is typically diagnosed using imaging tests such as magnetic resonance imaging (MRI) or Computed Tomography (CT) scans. Aortitis is an inflammation of the aorta, leading to a range of symptoms such as fever, weight loss, fatigue, and chest pain. In severe cases, aortic aneurysms or aortic dissection can occur, which can be life-threatening.

Multiple reports have demonstrated the presence of abnormal pro-inflammatory cytokine production in large-vessel vasculitis patients, particularly those with GCA, including interleukin-1 (IL-1), IL-6, IL-18, tumor necrosis factor-α (TNF-α), and interferon-γ, by T lymphocytes and macrophages. IL-6 has been implicated as a crucial cytokine in the pathogenesis of aortitis and targeting its signaling has shown promising results in treating the condition. IL-6 inhibitors such as tocilizumab have been found to effectively reduce disease activity and improve clinical outcomes in GCA patients.

The GIACTA study (GiAnt cell arteritis roActemra (tocilizumab) study) was a randomized, double-blind, placebo-controlled trial that evaluated the efficacy and safety of tocilizumab in the treatment of GCA. The study included 251 patients with newly diagnosed or relapsing GCA and found that treatment with tocilizumab significantly increased the proportion of patients who achieved sustained remission from GCA at 52 weeks, compared to placebo. Additionally, tocilizumab was associated with a lower incidence of disease flares and a reduced need for glucocorticoid therapy.

Following the positive results of the GIACTA study, tocilizumab was approved for the treatment of GCA in adults with active disease, including aortitis, who have not responded to glucocorticoids, or for whom glucocorticoid therapy is not appropriate, by regulatory agencies around the world, including the US Food and Drug Administration and the European Medicines Agency.

However, the efficacy of IL-6 inhibitors on aorta inflammation as assessed by modern and powerful imaging techniques has never been specifically studied in GCA.

This observational study will provide important informations on the impact of Tyenne® (tocilizumab) associated with short term low dose steroids on clinical manifestations and vessel inflammation and damage in aortitis of GCA.

DETAILED DESCRIPTION:
This is a prospective, observational study involving patients with active aortitis related to GCA.

After verification of the inclusion and exclusion criteria, and signature of the consent form, patients are included in the study. Patients will be followed and managed according to standard of care (visits and exams).

Oral corticosteroids must be at a stable dose for at least 2 weeks prior to the first administration of study drug at D0.

* All patients will receive oral prednisone ≥ 10 mg/day (or oral corticosteroid equivalent) with a maximum of 60 mg/day of prednisone or equivalent.
* A standardized prednisone reduction schedule (see below) will be applied to all groups as long as the disease is inactive, until prednisone is stopped. The aim is to taper off corticosteroids within eight weeks.
* At D0, MSB11456 / 1 injection S/C weekly will be initiated
* Blood samples will be taken every month up to week 52 for assessment of toxicity and inflammation markers.
* Assessment of adverse events will be done routinely at weeks 12, 24, 36, 52 and 104.
* Clinical evaluation will be performed routinely at weeks 12, 24, 36, 52 and 104.
* Targeted imaging studies (angio-CT) will be performed routinely at 6, 12 and 24 months after the start of treatment and if new symptoms appear.
* FDG Pet scan will be performed routinely at 6, 12 and 24 months after the start of treatment
* Angio-CT and FDG Pet scan will be proofread centrally. A standardized prednisone reduction schedule (see below) will be applied to all patients as long as the disease is inactive, until prednisone is stopped :

Baseline prednisone dose Corresponding dose (mg/day) at each week

CG(mg/d) ____60_____50_____40_____30_____25_____20_____15____10____7.5 (at baseline)

60__________W0

50__________W1____W0

40__________W2____W1____W0

30__________W3____W2____W1____W0

25___________ - ____W3____W2____W1____W0

20__________W4____W4____W3____W2____W1____W0

15__________W5____W5____W4____W3____W2____W1____W0

10__________W6____W6____W5____W4____W3____W2____W2____W0

7.5__________ - _____ - ______ - _____W5____W4____W3____W3____W1____W0

5 ___________W7____W7____W6____W6____W5____W4____W4____W2____W2

0 ___________W8____W8____W7____W7____W6____W6____W5____W4____W4

Sample size:

The investigators anticipated a remission rate of 70% at weel 24 based on pooled data from Viliger et al (1) and Stone et al (2). Viliger et al reported 85% of GCA remission at week 12 and week 52 with tocilizumab(1). Stone et al reported 56% of remission of GCA at week 52 under tocilizumab weekly with less than 10% of relpases between week 24 and week 52 (2). A total of 80 patients will ensure estimating the 24-week remission rate with a precision of +/- 11% using an exact 95% confidence intervalgiven the expected 70% remission rate.

Statistical analysis:

Descriptive analyses will be performed with counts and percent for discrete variables and median and interquartile range for continuous variables. The primary endpoint will be described with the 24-week remission proportion point estimate and its exact 95% confidence interval (95%CI) (Clopper Pearson). Secondary endpoints will be described using a similar approach for binary endpoints,continuous endpoints will be decsribed unsing median (IQR) and also mean (SD) with approximate Gaussian 95%CI for the mean.Kaplan Meier estimator or cumulative incidence estimates allowing competing risks when appropriate (i.e. treatment discontinuation due to toxicity), will be used for right-ecensored time to event variables, with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Signed informed consent
* Affiliation with the French national social security system
* Adequate and effective contraceptive measures
* For women of childbearing age, a negative serum pregnancy test.
* Diagnosis of GCA according to 2022 ACR/EULAR criteria
* Active newly diagnosed or relapsing Aortitis related to GCA proved by imaging (Tep-scan, angio-CT or magnetic resonance imaging angiography)
* No neoplasia
* No contraindication to Tocilizumab

Exclusion Criteria:

* Pregnancy or breastfeeding ;
* History of severe immunosuppression, HIV or HBsAg positive
* Non response or intolerance to previous therapy with tocilizumab
* Positive QuantiFERON test result (QFT-TBGIn-Tube)
* Have received live vaccines within 3 months prior to the start of the trial
* History of malignancy in the last 5 years
* Severe renal impairment (creatinine clearance <30mL/min/1.73m²)
* Liver dysfunction defined as aspartate transaminase (AST) or alanine transaminase (ALT) levels ≥ 5 at the upper limit of normal
* Blood count abnormality:

  * Platelet count < 50 x 10.3/mm3
  * Neutropenia < 1000/mm3
  * Hemoglobin < 8 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with active aortitis associated with GCA, requiring treatment with Tocilizumab biosimilar within the scope of its market authorization (standard of care)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2028-03-27 (Estimated)

PRIMARY OUTCOMES:
To evaluate the proportion of patients with remission of GCA | week 24
  Proportion of patients with remission of GCA at week 24. EULAR consensus definitions for remission in GCA and other types of LVV is defined as the absence of all clinical signs and symptoms attributable to active LVV, normalization of ESR and CRP values, and no evidence of progressive aortic damage at angio CT and Tep FDG.

SECONDARY OUTCOMES:
To assess the cumulative incidence of relapse | Weeks 12, 24, 36 , 52 and 104
  Cumulative incidence of relapse
To assess the proportion of GCA in remission (according to EULAR consensus definitions) after treatment start | Weeks 12, 24, 36 , 52 and 104
  Proportion of GCA in remission according to EULAR consensus definitions) after treatment start
To assess the cumulative dose of prednisone | Weeks 12, 24, 36, 52 and 104
  Cumulative prednisone dose
To assess the cumulative incidence of severe adverse events | Weeks 12, 24, 36, 52 and 104
  * Glucocorticoid Toxicity Index (GTI) at Weeks 24, 52 and 104;
  * Cumulative incidence of severe adverse events at Weeks 12, 24, 36 , 52 and 104, defined as those of grades III, IV or V, according to the Common Terminology Criteria for Adverse Events (CTCAE);
To assess the proportion of radiological vascular progression | Weeks 12, 24, 36 , 52 and 104
  Proportion of radiological vascular progression defined by :
  * new vascular lesions detected in CTA
  * new vascular lesions detected in Tep-scan
To assess the cumulative incidence of vascular revascularization procedures | Weeks 24, 52 and 104
  Cumulative incidence of vascular revascularization procedures needs (either endovascular or surgical) required due to inflammatory vascular activity

CONTACTS AND LOCATIONS:
Locations (1):
- Département de Medecine interne et d'immunologie clinique - hôpital La Pitié Salpetrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Villiger PM, Adler S, Kuchen S, Wermelinger F, Dan D, Fiege V, Butikofer L, Seitz M, Reichenbach S. Tocilizumab for induction and maintenance of remission in giant cell arteritis: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet. 2016 May 7;387(10031):1921-7. doi: 10.1016/S0140-6736(16)00560-2. Epub 2016 Mar 4. PMID 26952547
- [Result] Stone JH, Tuckwell K, Dimonaco S, Klearman M, Aringer M, Blockmans D, Brouwer E, Cid MC, Dasgupta B, Rech J, Salvarani C, Schett G, Schulze-Koops H, Spiera R, Unizony SH, Collinson N. Trial of Tocilizumab in Giant-Cell Arteritis. N Engl J Med. 2017 Jul 27;377(4):317-328. doi: 10.1056/NEJMoa1613849. PMID 28745999
- [Result] Hellmich B, Agueda A, Monti S, Buttgereit F, de Boysson H, Brouwer E, Cassie R, Cid MC, Dasgupta B, Dejaco C, Hatemi G, Hollinger N, Mahr A, Mollan SP, Mukhtyar C, Ponte C, Salvarani C, Sivakumar R, Tian X, Tomasson G, Turesson C, Schmidt W, Villiger PM, Watts R, Young C, Luqmani RA. 2018 Update of the EULAR recommendations for the management of large vessel vasculitis. Ann Rheum Dis. 2020 Jan;79(1):19-30. doi: 10.1136/annrheumdis-2019-215672. Epub 2019 Jul 3. PMID 31270110